CLINICAL TRIAL: NCT06219213
Title: Impact of a Daily Application of Serum and Cream Containing Glyceryl Eicosapentaenoate and Short-chain Fatty Acids on Skin Hydration: Exploratory Study (COS-PBP-01)
Brief Title: Glyceryl Eicosapentaenoate Based Topic Products As an Irritant-free Cream and Serum for Hydration of Sensitive Skin
Acronym: COS-PBP-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SCF Pharma (Industry)
Collaborators: Institut de recherche clinique du littoral (IRCL) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: COS-PBP-01
Record Dates: First submitted 2024-01-12; First posted 2024-01-23 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Skin Dryness
Keywords: Skin hydration; Skin inflammation; Eczema
MeSH Terms: conditions — Dermatitis; Eczema

STUDY DESIGN:
Intervention Model Description: The first eleven (11) subjects enrolled will be assigned to group A. Group B will follow with the eleven next subjets (subjects 12 to 22) and group C will complete the study with subjects 23 to 33. The pre-treatment state of subjects will serve as control for the effects observed following treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A: Cream of formulation A (Experimental): Daily application of glyceryl Eicosapentaenoate serum and glyceryl Eicosapentaenoate cream of formulation A on both targeted skin area. The skin areas must be clean and dry. Subjects may proceed with additional product applications if needed. However, for each additional application, both targeted areas must be treated with the Serum and the cream. Subjects must proceed with at least one application of products each day for 14 consecutive days.
  Interventions: Other: Glyceryl Eicosapentaenoate serum; Other: Glyceryl Eicosapentaenoate Cream A
- Group B: Cream of formulation B (Experimental): Daily application of glyceryl Eicosapentaenoate serum and glyceryl Eicosapentaenoate cream of formulation B on both targeted skin area. The skin areas must be clean and dry. Subjects may proceed with additional product applications if needed. However, for each additional application, both targeted areas must be treated with the Serum and the cream. Subjects must proceed with at least one application of products each day for 14 consecutive days.
  Interventions: Other: Glyceryl Eicosapentaenoate serum; Other: Glyceryl Eicosapentaenoate Cream B
- Group C: Cream of formulation C (Experimental): Daily application of glyceryl Eicosapentaenoate serum and glyceryl Eicosapentaenoate cream of formulation C on both targeted skin area. The skin areas must be clean and dry. Subjects may proceed with additional product applications if needed. However, for each additional application, both targeted areas must be treated with the Serum and the cream. Subjects must proceed with at least one application of products each day for 14 consecutive days.
  Interventions: Other: Glyceryl Eicosapentaenoate serum; Other: Glyceryl Eicosapentaenoate Cream C

INTERVENTIONS:
Other: Glyceryl Eicosapentaenoate serum — Daily application of serum on both targeted skin areas for 14 consecutive days. Serum must be applied before the Cream on clean skin.
Other: Glyceryl Eicosapentaenoate Cream A — Daily application of cream on both targeted skin areas for 14 consecutive days. Cream must be applied after the serum.
  Arms: Group A: Cream of formulation A
Other: Glyceryl Eicosapentaenoate Cream B — Daily application of cream on both targeted skin areas for 14 consecutive days. Cream must be applied after the serum.
  Arms: Group B: Cream of formulation B
Other: Glyceryl Eicosapentaenoate Cream C — Daily application of cream on both targeted skin areas for 14 consecutive days. Cream must be applied after the serum.
  Arms: Group C: Cream of formulation C

SUMMARY:
This exploratory study aims to verify the hydrating potential as well as the possible irritant effects of a 14-day hydrating treatment consisting of daily application of serum and cream to the skin of two dry targeted areas. Thirty-three (33) subjects will be enrolled in this study and will be divided into three different treatment groups of 11 subjects each. Apart from the formulation of the cream which varies between the three groups, the subjects will receive the same serum and adhere to the same study plan for fourteen days. Each subject's baseline condition before treatment will serve as a control for effects observed after treatment on targeted areas.

DETAILED DESCRIPTION:
The aim of this study is to verify the moisturizing potential of three different creams containing glyceryl eicosapentaenoates when used as a moisturizing treatment combined with a glyceryl eicosapentaenoate serum. Thirty-three (33) subjects will be enrolled in this study and will be divided into three different treatment groups of 11 subjects each. Before the first treatment, research staff must identify two areas of skin for each subject, ideally with different appearances. The assigned treatment will be applied to the targeted areas which will be used to measure hydration and redness. Apart from the formulation of the cream which varies between the three groups, subjects will receive the same serum and adhere to the same study plan. Subjects will be asked to apply the serum and cream to the targeted clean areas at least once a day, every day, for a period of fourteen (14) days. The baseline state before treatment will serve as a control for the effects observed after treatment on the targeted areas. The targeted areas will be used to measure hydration and redness:

1. Measure the skin hydration rate in the two selected areas by corneometry at the start of the study (pre-treatment), as well as after one (1) and two (2) weeks of treatment (at visits 2 and 3).
2. Measure the redness of the skin in the two selected areas by mexametry at the start of the study (pre-treatment), as well as after one (1) and two (2) weeks of treatment (at visits 2 and 3).

This study will help to evaluate and refine the treatment plan (frequency of application, duration of treatment, etc.) for future research projects with the same products. It will also assess the safety of the different formulations of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Participant aged between 18 and 65 years old.
* Participant who reports having dry skin.
* Available for the entire duration of the study and willing to participate based on the information provided in the informed consent form duly read and signed by the latter.
* Participant not presenting intellectual problems likely to limit the validity of consent to participate in the study and compliance with protocol requirements, having the ability to cooperate adequately, understand and observe the instructions of research staff.

Exclusion Criteria:

* Participant with a skin disease diagnosed by their treating physician and who requires drug treatment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2025-07-24 (Estimated); Study Completion 2025-08-07 (Estimated)

PRIMARY OUTCOMES:
Measure of Hydration | 2 weeks
  For each subject in every group, skin hydration will be measured by corneometry at baseline (visit 1/ pre-treatment) and after one (1) week of treatment (visit 2) and two (2) weeks of treatment (visit 3). Only the targeted treated areas will be used for the measure of hydration.
Measure of skin redness | 2 weeks
  For each subject in every group, skin redness will be measured by mexametry at baseline (visit 1/ pre-treatment) and after one (1) week of treatment (visit 2) and two (2) weeks of treatment (visit 3). Only the targeted treated areas will be used for the measure of redness.

SECONDARY OUTCOMES:
Control of skin appearance and adverse events | 2 weeks
  At each study visit, every subjet will be questioned for any adverse effect observed on targeted (treated) areas. Photos of both targeted areas will also be taken for every subject at each study visit. No measure or quantification are planned for these photos. They will remain in the files as documentation and will only be used if an adverse event need investigation.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Fortin, Ph.D, Principal Investigator — SCF Pharma
Locations (1):
- Institut de recherche clinique du littoral (IRCL), Rimouski, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The results of this research are the private property of SCF Pharma. If you are interested in the results of this study, you can contact Dr Samuel Fortin for a summary starting in summer 2025.

REFERENCES:
- [Background] Purnamawati S, Indrastuti N, Danarti R, Saefudin T. The Role of Moisturizers in Addressing Various Kinds of Dermatitis: A Review. Clin Med Res. 2017 Dec;15(3-4):75-87. doi: 10.3121/cmr.2017.1363. Epub 2017 Dec 11. PMID 29229630
- [Background] Hsu CK, Cheng NY, Yang CC, Yen YY, Tseng SH. Investigating the clinical implication of corneometer and mexameter readings towards objective, efficient evaluation of psoriasis vulgaris severity. Sci Rep. 2022 May 6;12(1):7469. doi: 10.1038/s41598-022-11573-2. PMID 35523995